CLINICAL TRIAL: NCT04717336
Title: Genomics, Environmental Factors and Social Determinants of Cardiovascular Disease in African-Americans Study(GENE-FORECAST): Sodium Intervention Trial (SIT)/GENE-FORECAST SIT
Brief Title: Genomics, Environmental Factors and Social Determinants of Cardiovascular Disease in African Americans Study (GENE-FORECAST): Sodium Intervention Trial (SIT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 10000070; 000070-H
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Results first posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2024-07-23

CONDITIONS: Cardiovascular Disease
Keywords: African American; Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Sodium Chloride then Placebo (Experimental): Participant will take Sodium Chloride at 3 pills per day for a total of 3 grams for two weeks, followed by a wash-out period for three-weeks, then ending with a cross-over to the Placebo at 3 pills per day for a total of 3 grams for two weeks.
  Interventions: Other: Sodium Chloride; Other: Placebo
- Cohort 2: Placebo then Sodium Chloride (Experimental): Participant will take Placebo at 3 pills per day for a total of 3 grams for two weeks, followed by a wash-out period for three-weeks, then ending with a cross-over to the Sodium Chloride at 3 pills per day for a total of 3 grams for two weeks.
  Interventions: Other: Sodium Chloride; Other: Placebo

INTERVENTIONS:
Other: Sodium Chloride — It is well established that increased dietary sodium can predispose to an increase in blood pressure; particularly in salt-sensitive individuals. Seeking to test the hypothesis that changes in dietary sodium intake are sufficient to influence the composition of the gut microbiome in association with sodium-induced changes in vascular function, epigenome, transcriptome and blood pressure in African Americans.
  Other Names: salt treatment
Other: Placebo — placebo capsules

SUMMARY:
Background:

Hypertension is a risk factor for heart disease. Low-sodium diets rich in fruits, vegetables, and other healthy foods are a good way to reduce blood pressure in people with hypertension. Researchers want to learn more about why African Americans seem to have the greatest benefit from certain dietary interventions.

Objective:

To better understand the body's response to adding more salt to the diet.

Eligibility:

U.S.-born African American adults ages 21 to 65 who are in good general health and took part in the GENE-FORECAST.

Design:

Participants will be screened with a medical history and physical exam. If needed, they will take a pregnancy test. These tests will be repeated during the study.

Each day for 2 weeks, participants will take 3 capsules that contain either placebo or salt. Then they will take no pills for 3 weeks. Then they will take placebo or salt capsules for 2 more weeks.

Participants will talk about the foods and drinks they have consumed over the past 24 hours. They will take a survey about their physical activity and sleep.

Participants will complete taste tasks to obtain their responses to sweetness or saltiness. Sucrose and salt detection thresholds and preferences will be assessed.

Participants will give blood and urine samples. Saliva samples will be collected from their mouth by passive drool or by spitting into a sterile tube. Skin samples will be collected from behind their ears and the inner part of their elbow, using sterile swabs. Participants will get kits to collect stool samples at home.

Participants will have 4 study visits over 7 weeks.

DETAILED DESCRIPTION:
The objective of this study is to implement a sodium intervention investigation to assess the effect of increased dietary sodium intake on changes in blood pressure, vascular function, microbiome, whole blood epigenome, whole blood and urine transcriptome as outcome measures. The study design will include a double-blind, cross-over treatment/placebo trial among African Americans GENE-FORECAST participants with normal blood pressure and will last 7 weeks. It is hypothesized that exposure to increased dietary sodium will affect blood pressure, whole blood epigenome, whole blood and urine transcriptome, vascular function, microbiome and blood pressure.

ELIGIBILITY:
* INCLUSION CRITERIA:

African American men and women who are former GENE-FORECAST participants between 21 and 65 years of age. This criterion is inclusive of self-identified AA of both Hispanic, Latino and non-Hispanic, Latino ethnicities. Normotensive participants with systolic blood pressure (SBP) <140 mm Hg and diastolic blood pressure (DBP) <90 mm Hg and the absence of a history of prior diagnosis of hypertension.

-Willingness and ability to participate in study procedures.

EXCLUSION CRITERIA:

* Individuals who are pregnant or breast-feeding.
* Individuals with high blood pressure or a history of hypertension.
* Individuals with a history of myocardial infarction, stroke, heart failure, diabetes, chronic liver or kidney diseases.
* Individuals who are taking antihypertensive, antidepressants, antidiabetic and antibiotic medications.
* Individuals currently participating in another NIH protocol.
* Individuals unable to provide informed consent.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amadou Gaye, PhD, Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000070-HG.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Sodium Chloride Then Placebo: Participant will take Sodium Chloride at 3 pills per day for a total of 3 grams for two weeks, followed by a wash-out period for three-weeks, then ending with a cross-over to the Placebo at 3 pills per day for a total of 3 grams for two weeks.
- Placebo Then Sodium Chloride: Participant will take Placebo at 3 pills per day for a total of 3 grams for two weeks, followed by a wash-out period for three-weeks, then ending with a cross-over to the Sodium Chloride at 3 pills per day for a total of 3 grams for two weeks.
Period: Period 1: Baseline to Week 2
Arm/Group | Sodium Chloride Then Placebo | Placebo Then Sodium Chloride
Started | 20 | 16
Completed | 18 | 14
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2
Period: Washout: Week 2 to Week 5
Arm/Group | Sodium Chloride Then Placebo | Placebo Then Sodium Chloride
Started | 18 | 14
Completed | 16 | 12
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2
Period: Period 2: Week 5 to Week 7
Arm/Group | Sodium Chloride Then Placebo | Placebo Then Sodium Chloride
Started | 16 | 12
Completed | 16 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sodium Chloride Then Placebo | Placebo Then Sodium Chloride | Total
Number analyzed (Participants) | 20 | 16 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 16 | 36
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 18 | 15 | 33
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 16 | 36
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 16 | 36

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Vascular Function Measured by Pulse Wave Velocity
Description: Mean change in vascular function was measured by Pulse Wave Velocity (PWV) using the SphygmoCor XCEL. PWV was determined by recording the pulse waves of the carotid and femoral arteries and calculating the ratio of the distance between the pulse measuring sites to the time delay between the carotid and femoral pulse waves. The distance was measured with a non-stretchable tape from the suprasternal notch to the carotid site and from the suprasternal notch to the femoral site. The former distance was subtracted from the latter and used in the calculation of PWV. High PWV is directly associated with increased arterial stiffness, reflecting reduced elasticity of the arterial walls.
Time Frame: Baseline, Week 2, Week 5 and Week 7
Population: Analysis includes only those participants that completed the Pulse Wave Velocity at every visit (n=23).
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Sodium Chloride Then Placebo | Placebo Then Sodium Chloride
Number analyzed (Participants) | 13 | 10
m/s
  Baseline | 7.08 (1.50) | 7.13 (0.81)
  Week 2 | 7.34 (0.88) | 7.07 (0.96)
  Week 5 | 6.88 (1.06) | 6.86 (1.30)
  Week 7 | 7.03 (1.27) | 6.70 (0.95)
Statistical Analysis 1: Comparison: Sodium Chloride Then Placebo vs Placebo Then Sodium Chloride; The aim of this analysis is to test whether there is a statistically significant difference in Pulse Wave Velocity when participants are on sodium chloride vs. placebo, regardless of period; Test type: Superiority; p = 0.98, Paired T-Test; A paired t-test was applied across both periods because this is a cross-over study where each participant serves at their own control; Mean of Paired Differences = 0.002, 95% CI 2-sided [-0.22 to 0.23]

ADVERSE EVENTS:
Time Frame: 7 weeks
Groups:
- Sodium Chloride: Participant will take Sodium Chloride at 3 pills per day for a total of 3 grams for two weeks.
- Placebo: Participant will take Placebo at 3 pills per day for a total of 3 grams for two weeks.
- Wash-Out Period: Participants do not take any study intervention for this washout period.
Arm/Group | Sodium Chloride | Placebo | Wash-Out Period
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 1/32 | 1/32 | 0/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Chloride (N=32) | Placebo (N=32) | Wash-Out Period (N=32)
Hives (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-29): https://cdn.clinicaltrials.gov/large-docs/36/NCT04717336/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-12): https://cdn.clinicaltrials.gov/large-docs/36/NCT04717336/ICF_001.pdf